CLINICAL TRIAL: NCT07153497
Title: A Randomized Phase 2 Trial of Olutasidenib-Based Therapies in Patients With Newly Diagnosed IDH1-Mutant Myeloid Malignancies: A MyeloMATCH Substudy
Brief Title: Testing the Use of an IDH1 Inhibitor, Olutasidenib, in Acute Myeloid Leukemia Added to ASTX727 and Venetoclax; in High-Risk MDS Added to ASTX727; and Alone in Low Risk MDS (A MyeloMATCH Treatment Substudy)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-06184; NCI-2025-06184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1OA-MDS-A05 (Other: Alliance for Clinical Trials in Oncology); MM1OA-MDS-A05 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2025-09-03; First posted 2025-09-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; olutasidenib; venetoclax

STUDY DESIGN:
Intervention Model Description: Cohort A: Randomization to Arm 1 or Arm 2; Cohort B: Randomization to Arm 3 or Arm 4; Cohort C: Assignment to single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A, Arm 1 (ASTX727, venetoclax) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Cohort A, Arm 2 (ASTX727, venetoclax, olutasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle, venetoclax PO QD on days 1-28 of each cycle, and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Olutasidenib; Drug: Venetoclax
- Cohort B, Arm 3 (ASTX727, olutasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Olutasidenib
- Cohort B, Arm 4 (ASTX727) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients without CR after cycle 6 may then cross-over to Arm 3. Patients with CR, as well as patients without CR but deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine
- Cohort C (olutasidenib) (Experimental): Patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Olutasidenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
  Arms: Cohort A, Arm 1 (ASTX727, venetoclax); Cohort A, Arm 2 (ASTX727, venetoclax, olutasidenib); Cohort B, Arm 3 (ASTX727, olutasidenib); Cohort B, Arm 4 (ASTX727)
Drug: Olutasidenib — Given PO
  Other Names: FT 2102; FT-2102; FT2102; IDH1-R132 Inhibitor FT-2102; Rezlidhia
  Arms: Cohort A, Arm 2 (ASTX727, venetoclax, olutasidenib); Cohort B, Arm 3 (ASTX727, olutasidenib); Cohort C (olutasidenib)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Cohort A, Arm 1 (ASTX727, venetoclax); Cohort A, Arm 2 (ASTX727, venetoclax, olutasidenib)

SUMMARY:
This phase II MyeloMATCH treatment substudy tests the addition of olutasidenib to usual treatment in patients with higher-risk myelodysplastic syndrome (MDS) or patients with acute myeloid leukemia (AML) with a mutation in the IDH1 gene. Olutasidenib blocks the protein made by the mutated IDH1 gene. Blocking this protein may help keep cancer cells from growing. For patients with MDS, olutasidenib will be added to decitabine-cedazuridine (also called ASTX727). Decitabine is in a class of medications called hypomethylating agents and is the standard treatment for MDS. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. The cedazuridine makes it possible to take the decitabine by mouth. Adding olutasidenib to the usual treatment for MDS (ASTX727) may increase the likelihood of going into remission. For patients with AML, olutasidenib and ASTX727 will be combined with venetoclax, a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. Venetoclax may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Adding olutasidenib to the usual treatment for AML (ASTX727 and venetoclax) may increase the likelihood of going into remission. For low risk MDS, the substudy tests whether giving olutasidenib alone helps improve blood counts.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of minimal residual disease (MRD)-negative composite complete response (CRc) (CR + CR with partial hematological recovery [CRh] + CR with incomplete bone marrow recovery [CRi]), based on multiparametric flow cytometry (MFC), in older adults with IDH1-mutant acute myeloid leukemia (AML) treated with decitabine and cedazuridine (ASTX727), venetoclax (VEN), and olutasidenib compared to ASTX727 plus VEN, within 4 cycles of treatment. (Cohort A: IDH1-mutant AML) II. To assess the CR rate (including CR equivalent), using the modified International Working Group (IWG) 2023 response criteria, for patients with IDH1-mutant high-risk (HR)-MDS treated with ASTX727 plus olutasidenib compared to ASTX727 alone. (Cohort B: IDH1-mutant HR-MDS) III. To assess the rate of hematologic improvement (HI), using the IWG 2018 response criteria, for patients with IDH1-mutant low risk (LR)-MDS treated with olutasidenib. (Cohort C: IDH1-mutant LR-MDS)

SECONDARY OBJECTIVES:

I. To compare the rate of CR and composite CR (CR, CRh, CRi) by treatment arm. (Cohort A: IDH1-mutant AML) II. To compare the rate and duration of transfusion independence by treatment arm. (Cohort A: IDH1-mutant AML) III. To compare the event-free survival (EFS), cumulative incidence of relapse (CIR), early mortality, and overall survival (OS) by treatment arm. (Cohort A: IDH1-mutant AML) IV. To estimate the frequency and severity of toxicities by treatment arm. (Cohort A: IDH1-mutant AML) V. To compare the clearance of IDH1 mutation in bone marrow by treatment arm. (Cohort A: IDH1-mutant AML) VI. To compare the correlation between MRD clearance (including MFC and molecular MRD) and survival (including OS and EFS) by treatment arm. (Cohort A: IDH1-mutant AML) VII. To compare the rate of composite CR (CR [or CR equivalent] + CR with lesser hematological recovery [CRL] [CR with unilineage recovery (CRuni), CR with bilineage recovery (CRbi)] + CRh) using the modified IWG 2023 response criteria for patients with IDH1-mutant HR-MDS treated with ASTX727 plus olutasidenib compared to ASTX727 alone. (Cohort B: IDH1-mutant HR-MDS) VIII. To compare the overall response rate (ORR; defined as CR [or CR equivalent] + partial response [PR] + CRL [CRuni, CRbi] + CRh + HI) using the modified IWG 2023 response criteria for each treatment arm. (Cohort B: IDH1-mutant HR-MDS) IX. To compare the rate and duration of transfusion independence by treatment arm. (Cohort B: IDH1-mutant HR-MDS) X. To compare the time to response and duration of response (DoR) by treatment arm. (Cohort B: IDH1-mutant HR-MDS) XI. To compare the EFS and OS of patients by treatment arm. (Cohort B: IDH1-mutant HR-MDS) XII. To estimate the frequency and severity of toxicities by treatment arm. (Cohort B: IDH1-mutant HR-MDS) XIII. To compare the rate of patients bridged to allogeneic stem cell transplantation (allo-SCT) by treatment arm. (Cohort B: IDH1-mutant HR-MDS) XIV. To compare the clearance of IDH1 mutation, in bone marrow by treatment arm and correlation with survival (including OS and EFS) (Cohort B: IDH1-mutant HR-MDS) XV. To compare ORR, EFS, and OS by treatment arm stratified by the Molecular International Prognostic Scoring System for Myelodysplastic Syndromes (IPSS-M) prognostic scoring system. (Cohort B: IDH1-mutant HR-MDS) XVI. To estimate the rate of CR, median EFS, and median OS in patients who do not achieve CR with ASTX727 monotherapy, who are treated with the combination of ASTX727 plus olutasidenib. (Cohort B: IDH1-mutant HR-MDS) XVII. In patients with red blood cell transfusion-dependent (RBC-TD) anemia: To assess the rate of 8-week and 24-week red blood cell (RBC) transfusion independence (RBC-TI) with olutasidenib, time to RBC-TI, rate of transformation to AML and rate of 1-year RBC-TI. (Cohort C: IDH1-mutant LR-MDS) XVIII. To estimate the frequency and severity of toxicities with olutasidenib. (Cohort C: IDH1-mutant LR-MDS) XIX. To estimate rate of cytogenetic response (in patients with baseline cytogenetic abnormalities) and IDH1 mutational clearance with olutasidenib and correlation with rate of HI. (Cohort C: IDH1-mutant LR-MDS)

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT A: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ASTX727 orally (PO) once daily (QD) on days 1-5 of each cycle and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

ARM 2: Patients receive ASTX727 PO QD on days 1-5 of each cycle, venetoclax PO QD on days 1-28 of each cycle, and olutasidenib PO twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

COHORT B: Patients are randomized to 1 of 2 arms.

ARM 3: Patients receive ASTX727 PO QD on days 1-5 of each cycle and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

ARM 4: Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients without CR after cycle 6 may then cross-over to Arm 3. Patients with CR, as well as patients without CR but deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

COHORT C: Patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be enrolled on the MYELOMATCH Master Screening and Reassessment Protocol (MSRP), determined to have an IDH1-R132 mutation and assigned to this trial via MATCHBox
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1):
* Documentation of IDH1 mutated MDS or AML
* COHORT A: Age ≥ 60 years or adults ˂ 60 and ≥ 18 who in the opinion of the treating physician are not candidates for intensive, cytarabine-based induction based on clinical status (i.e., performance status), organ dysfunction, or disease biology with a morphologically confirmed diagnosis of AML with ≥ 20% myeloblasts in the bone marrow or peripheral blood
* COHORT B: Age ≥ 18 years with treatment-naïve HR-MDS with an IPSS-R score ≥ 4.0 at time of enrollment
* COHORT C: Age ≥ 18 years with LR-MDS with an IPSS-R score ≤ 3.5 at time of enrollment and either:

  * RBC-TD anemia (≥ 2 units/8 weeks in the 16 weeks prior to registration) who have failed or are ineligible to erythropoiesis-stimulating agents (ESA) therapy
  * Presence of either neutropenia (< 1 x 10^9/L) or thrombocytopenia (< 100 x 10^9/L) for use as frontline therapy or after failure of prior therapies, including growth factors. Patient must be hypomethylating agent (HMA)-naïve
* No prior therapy excluding:

  * Cohort A: hydroxyurea and all-trans retinoic acid (ATRA) for AML
  * Cohort B: ESAs (erythropoiesis-stimulating agents) and/or TGF-β inhibitors for HR-MDS
  * Cohort C: ESAs (erythropoiesis-stimulating agents, TGF-β inhibitors, telomerase inhibitors, and/or G-CSF for LR-MDS)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 3
* Creatinine clearance ≥ 30 mL/min (using the Cockcroft-Gault equation)
* Total bilirubin ≤ 3 x upper limit of normal (ULN)

  * Unless the increase is due to Gilbert's disease as determined per physician discretion/institutional practice
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x upper limit of normal (ULN)
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effect on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test must be done ≤ 7 days prior to registration. (Cohorts B and C only)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. A corrected QT interval < 480 msec (calculated using the Fridericia's formula [QTcF]) excluding patients with a right bundle branch block (RBBB) after approval of the principal investigator (PI)
* No known medical condition causing an inability to swallow, tolerate oral medications and must have no known malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or small bowel resection) that may significantly alter the absorption of the study drugs
* RE-REGISTRATION ELIGIBILITY CRITERIA FOR COHORT B, ARM 3 (STEP 2): Patients on the ASTX727 monotherapy arm (Cohort B-Arm 3) that do not achieve a CR (complete response), CRL (CR with limited count recovery), or CRh (CR with partial count recovery) after completing 6 cycles of study treatment
* RE-REGISTRATION ELIGIBILITY CRITERIA FOR COHORT B, ARM 3 (STEP 2): ECOG Performance Status ≤ 3
* RE-REGISTRATION ELIGIBILITY CRITERIA FOR COHORT B, ARM 3 (STEP 2): Creatinine clearance ≥ 30 mL/min (using the Cockcroft-Gault equation)
* RE-REGISTRATION ELIGIBILITY CRITERIA FOR COHORT B, ARM 3 (STEP 2): Total bilirubin ≤ 3 x upper limit of normal (ULN)

  * Unless the increase is due to Gilbert's disease as determined per physician discretion/institutional practice
* RE-REGISTRATION ELIGIBILITY CRITERIA FOR COHORT B, ARM 3 (STEP 2): AST (SGOT)/ALT (SGPT) ≤ 3 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-05-27 (Estimated); Primary Completion 2030-04-26 (Estimated); Study Completion 2030-04-26 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD)-negative complete response (CR) + CR with partial hematological recovery (CRh) + CR with incomplete bone marrow recovery (CRi) (Cohort A) | Up to 4 cycles post randomization (Cycles = 28 days)
  Will compare the MRD-negative composite complete response (CRc) rate between the two treatment arms to determine if older adults with IDH1-mutant acute myeloid leukemia (AML) treated with the triplet ASTX727, venetoclax (VEN), and olutasidenib have a statistically significantly higher MRD-negative CRc rate than patients treated with the doublet ASTX727 and VEN. CRc will be determined based on multiparametric flow cytometry.
Rate of CR (Cohort B) | Up to 6 cycles post randomization (Cycles = 28 days)
  Will include CR equivalent. Will compare the CR rate between the two treatment arms to determine if patients with IDH1-mutant higher-risk-myelodysplastic syndrome (MDS) treated with ASTX727 plus olutasidenib have a statistically significantly higher CR rate than those treated with ASTX727 alone. Complete response will be determined using the modified International Working Group (IWG) 2023 response criteria.
Rate of hematologic improvement (HI) (Cohort C) | Up to 6 cycles post randomization (Cycles = 28 days)
  Will be determined using the IWG 2018 response criteria for patients with IDH1-mutant low risk-MDS treated with olutasidenib.

SECONDARY OUTCOMES:
CR and CRc (Cohort A) | Up to 5 years
  CRc will be defined as CR, CRh, or CRi. Both the CR rate and the composite CR rate will be determined for each treatment arm. The difference in rate between the two arms will be provided along with a 95% confidence interval.
Transfusion independence (Cohorts A) | Up to 5 years
  Will report the difference in rate of transfusion independence between the two treatment arms along with a 95% confidence interval. Additionally, will report the duration of transfusion independence, defined as the time from randomization to transfusion dependence, with the corresponding hazard ratio and Kaplan Meier curve.
Event-free survival (EFS) (Cohort A) | From randomization until either a failure to achieve a CRc after four cycles of treatment, relapse, or death due to any cause, assessed up to 5 years
  Sensitivity analyses will be conducted to evaluate different definitions in EFS, e.g., patients who failed to achieve a CR, CRh, or Cri after four cycles of treatment will be censored at the time of randomization. Will utilize the methods of Kaplan-Meier as well as Cox regression models to evaluate these time-to-event outcomes.
Cumulative incidence of relapse (Cohort A) | From which a patient achieves a CR to the time of relapse, assessed up to 5 years
  A cumulative incidence function will be created and a cause-specific hazard approach will be utilized with the event of interest being relapse and the competing risk being death.
Early mortality (Cohort A) | Up to 30 and 60 days
  Will be calculated as binomial distribution with corresponding 95% confidence intervals.
Overall survival (OS) (Cohort A) | From randomization to the time of death due to any cause, assessed up to 5 years
  Will utilize the methods of Kaplan-Meier as well as Cox regression models to evaluate time-to-event outcomes.
Incidence of adverse events (Cohort A, B, and C) | Up to 5 years
  As per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. In addition, will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The incidence of severe (grade 3+) adverse events or toxicities will be described for each treatment arm, but will also be compared between the arms. Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest between the treatment arms and will graphically assess differences in maximum grades observed for toxicities between the arms.
Composite CR (Cohort B) | Up to 5 years
  Will be defined as CR (or CR equivalent) + CR with lesser hematological recovery (CRL) (CR with unilineage recovery [CRuni], CR with bilineage recovery [CRbi]) + CRh, which will be determined by the IWG 2023 response criteria. The composite CR rate will be determined for each treatment arm. The difference in rate between the two arms will be provided along with a 95% confidence interval. Will also conduct an additional analysis to estimate the composite CR rate for patients who crossed over.
Overall response rate (ORR) (Cohort B) | Up to 5 years
  Will be defined as CR (or CR equivalent) + partial response + CRL (CRuni, CRbi) + CRh + hematologic improvement, which will be determined by the IWG 2023 response criteria. The overall response rate will be determined for each treatment arm. The difference in rate between the two arms will be provided along with a 95% confidence interval. Will also report results stratified by Molecular International Prognostic Scoring System for Myelodysplastic Syndromes (IPSS-M) score.
Transfusion independence (Cohort B) | Up to 5 years
  Will report the difference in rate of transfusion independence between the two treatment arms along with a 95% confidence interval. Additionally, will report the duration of transfusion independence, defined as the time from randomization to transfusion dependence, with the corresponding hazard ratio and Kaplan Meier curve.
Duration of response (Cohort B) | Up to 5 years
  Among patients who achieve a response (both composite response and ORR), duration of response will be defined as the time a patient first achieves a response until either progression or death. Only patients who achieve a response will be used for this analysis. Patients that withdraw early after achieving a response will be censored on their date of withdrawal. Patients who utilize alternative therapy won't be censored, but sensitivity analyses will be conducted. Will utilize the methods of Kaplan-Meier as well as Cox regression models to evaluate these time-to-event outcomes.
Event-free survival (EFS) (Cohort B) | From randomization until either a failure to achieve a CRc after four cycles of treatment, relapse, or death due to any cause, assessed up to 5 years
  Sensitivity analyses will be conducted to evaluate different definitions in EFS, e.g., patients who failed to achieve a CR, CRh, or Cri after four cycles of treatment will be censored at the time of randomization. Will utilize the methods of Kaplan-Meier as well as Cox regression models to evaluate these time-to-event outcomes. Additional planned analyses include reporting results stratified by IPSS-M score and estimating median EFS for patients that crossed over.
Overall survival (OS) (Cohort B) | From randomization to the time of death due to any cause, assessed up to 5 years
  Will utilize the methods of Kaplan-Meier as well as Cox regression models to evaluate time-to-event outcomes. Additional planned analyses include reporting results stratified by IPSS-M score and estimating median OS for patients that crossed over.
Allogeneic stem cell transplantation (Allo-SCT) bridge rate (Cohort B) | Up to 5 years
  Will report the difference in rate of rate of patients bridged to Allo-SCT between the two treatment arms along with a 95% confidence interval.
Transfusion independence (Cohort C) | Up to 5 years
  For patients with red blood cell transfusion-dependent (RBC-TD) anemia, will report the estimated rate of 8-week, 24-week, and 52-week RBC transfusion independence along with a 95% confidence interval. Additionally, will report the time to transfusion independence, defined as the time from randomization to transfusion independence, with the corresponding hazard ratio and Kaplan Meier curve.
Transformation to AML (Cohort C) | Up to 5 years
  For patients with RBC-TD anemia, will report the estimated rate of transformation to AML along with a 95% confidence interval.
Cytogenetic response (Cohort C) | Up to 5 years
  For patients with baseline cytogenetic abnormalities, will estimate the rate of cytogenetic response and provide a corresponding 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: John L Reagan, Principal Investigator — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm